CLINICAL TRIAL: NCT00642317
Title: Asian Youth and Tobacco Control Survey
Status: Completed | Type: Observational
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Other Study IDs: 2007-0901
Record Dates: First submitted 2008-03-19; First posted 2008-03-25 (Estimated); Last update posted 2012-08-01 (Estimated); Status verified 2012-07

CONDITIONS: Tobacco Use; Smoking
Keywords: Healthy Control; Tobacco Use; Tobacco Initiation; Smoking; Questionnaire; Survey
MeSH Terms: conditions — Tobacco Use; Smoking | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Asian Youth and Tobacco Control: Smoking Questionnaire for self-identified Chinese or Vietnamese participants.
  Interventions: Behavioral: Questionnaire

INTERVENTIONS:
Behavioral: Questionnaire — Questionnaire about tobacco and alcohol use, acculturation, and other related topics.
  Other Names: Survey

SUMMARY:
The overall goal of this study is to identify and understand the environmental characteristics associated with tobacco use and tobacco initiation among Asian American youth from primarily two communities: Chinese and Vietnamese. The specific aims of this study are twofold:

* To estimate the prevalence of smoking among Chinese and Vietnamese youth in the Houston area compared with non-Asian American communities.
* To study the relationship between environmental characteristics (both pro- and anti-tobacco) and tobacco initiation and use among Chinese and Vietnamese youth.
* To explore if degree of acculturation is related to tobacco initiation and use among Chinese and Vietnamese youth.

DETAILED DESCRIPTION:
This is a survey about health-related behaviors, risks, attitudes and acculturation. It includes questions about use of alcohol, tobacco, and other drugs; safety and violence; diet and physical activity; and youth programs and resources in your community. Your answers are completely anonymous, and your name will not appear anywhere on this survey or as part of this survey. Your parents will not see your responses.

ELIGIBILITY:
Inclusion Criteria:

* Self-identified male or female of Chinese or Vietnamese descent
* Age 12-17 years
* Living in the Greater Houston area
* Intellectual age of 7 or higher

Exclusion Criteria: None

Ages: 12 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Participants self-identified as having Chinese or Vietnamese descent.
Sampling Method: Non-Probability Sample
Enrollment: 617 (Actual)
Dates: Start 2008-03; Primary Completion 2009-01 (Actual); Study Completion 2009-01 (Actual)

PRIMARY OUTCOMES:
Prevalence Rates of smoking among Chinese and Vietnamese youth in the Houston area. | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Alex Prokhorov, MD, PhD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- U.T.M.D. Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: MD Anderson Cancer Center — http://www.mdanderson.org